CLINICAL TRIAL: NCT06005883
Title: The Prognosis After Surgical Resection in Patients With Hepatocellular Carcinoma Combined Portal Vein Tumor Thrombosis; Multicenter Retrospective Study
Brief Title: Surgical Outcome of HCC With Portal Vein Tumor Thrombosis on the Basis of Risk Scoring
Status: Completed | Type: Observational
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-03-065-003
Record Dates: First submitted 2023-08-08; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Thrombosis; Prognosis
Keywords: Hepatocellular carcinoma; portal vein tumor thrombosis; Prognosis; Hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this multicenter retrospective cohort study is to investigate the clinical outcomes and prognostic factors after hepatic resection in patients with HCC exhibiting PVTT, and to develop a prognostic index that can be helpful in determining the treatment strategy.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) frequently invades the surrounding liver vasculature, with portal vein tumor thrombosis (PVTT) being the most common form of macrovascular invasion. At the time of HCC diagnosis, PVTT is detected in approximately 10%-40% of patients and is associated with an extremely poor prognosis.

In most staging systems and guidelines, HCC with PVTT, regardless of the extent of the tumor, is classified as an advanced stage, and surgical resection is not recommended as the first-line treatment. Instead, consensus guidelines such as those from the American Association of Study of Liver Disease(AASLD), the Asian Pacific Association for the Study of Liver(APASL), and the European Association for the Study of Liver(EASL) recommend systemic and targeted therapy for these patients. Despite these recommendations, experienced liver centers in Asia have been attempting surgical resection for some patients with HCC exhibiting PVTT, and the outcomes are favorable in selected patients. However, most of the studies were conducted in only one center, had a small sample size, and obtained undesirable surgical treatment outcomes in most of the patients. Thus, surgical resection has not yet been widely accepted as an effective treatment for patients with HCC and PVTT. In addition, a prognostic index that can indicate which surgical resection is beneficial in comparison with nonsurgical treatment remains unestablished. A randomized controlled trial could be the best way to compare the outcomes of surgical resection and nonsurgical treatments, but it is difficult to conduct because of difficulties in ethical approval and allocation concealment. Therefore, adequate studies with large sample sizes are needed to clarify the benefits of surgical resection in patients with HCC and PVTT and the prognostic index, which can specify the criteria for surgical resection in these patients.

This study aimed to investigate the clinical outcomes and prognostic factors after hepatic resection in patients with HCC exhibiting PVTT, and to develop a prognostic index that can be helpful in determining the treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

The patients underwent liver resection for HCC with portal vein tumor thrombosis between Jan 2005 and Dec 2019 at 10 university-affiliated hospitals in South Korea.

Exclusion Criteria:

* Metastatic cancer & extrahepatic metastasis
* Intrahepatic cholangiocarcinoma
* Mixed type hepatocellular-cholangiocarcinoma
* Recurred hepatocellular carcinoma
* not available medical records.
* Child-Pugh classification B or C

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective multicenter study enrolled patients who underwent surgical resection of HCC with PVTT at 10 university-affiliated hospitals in Korea between January 2005 and December 2019. The institutional review board of each study center approved the study protocol (IRB No.:2022-03-065-003). The inclusion criteria were as follows: a) HCC with PVTT found on preoperative imaging and proven by postoperative histology whether it is viable; b) Child-Pugh class A liver function; c) no extrahepatic metastasis and concomitant malignant tumors other than HCC; d) no previous hepatic resection for HCC; and e) available medical records and/or imaging studies.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Death | From the date of surgery until the date of patient's death from any cause, whichever came first, assessed up to November 2021.
  Patient's death after surgical resection in HCC patients with portal vein tumor thrombosis
Recurrence of tumor | From the date of surgery until the date of HCC recurrence, whichever came first, assessed up to November 2021.
  HCC recurrence after surgical resection in HCC patients with portal vein tumor thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Keimyung university Dongsan Medical Center, Daegu, DalSeo-gu, South Korea